CLINICAL TRIAL: NCT07284745
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of KarXT + KarX-EC in Children and Adolescents (5 to 17 Years of Age) With Irritability Associated With Autism Spectrum Disorder
Brief Title: A Study of KarXT + KarX-EC for Treatment of Irritability in Children and Adolescents With Autism
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0044
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Irritability Associated With Autism Spectrum Disorder
Keywords: Cobenfy; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + KarX-EC Arm (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC
- Placebo (Placebo Comparator)
  Interventions: Drug: KarXT + KarX-EC Matching Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline/Trospium Chloride
  Arms: KarXT + KarX-EC Arm
Drug: KarX-EC — Specified dose on specified days
  Other Names: BMS-986519; Xanomeline Enteric-coated
  Arms: KarXT + KarX-EC Arm
Drug: KarXT + KarX-EC Matching Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess KarXT + KarX-EC for the treatment of irritability associated with autism in children and adolescents.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a confirmed diagnosis of ASD, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria, confirmed by the K-SADS-PL and must be experiencing symptoms of irritability.
* Participants must have ABC-I ≥18 (C18 on the Irritability subscale of the ABC-I) and CGIS specific to irritability ≥4, at screening and baseline (Day 1).

Exclusion Criteria

* Participants must not have a current primary DSM-5 diagnosis of bipolar disorder, including bipolar II disorder, schizophrenia, schizoaffective disorder, major depressive episode as determined by clinical instrument, or post-traumatic stress disorder (PTSD).
* Exception Include: Participants with comorbid ADHD, provided that attention deficit/hyperactivity disorder (ADHD) is not the primary disorder, the participant is adequately treated and based on the investigator judgment the disorder is clinically stable.
* Participants must not have history/presence of clinically significant disease or disorder that would jeopardize participant safety or validity of study results.
* Participants must not have a risk for suicidal behavior, and any clinically significant abnormal laboratory test.
* Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-07-05 (Estimated); Study Completion 2029-07-05 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Aberrant Behavior Checklist Irritability (ABC-I) Score at Week 8 | Week 8

SECONDARY OUTCOMES:
Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Score at Week 8 | Week 8
Number of Participants With ABC-I Response at Week 8 | Week 8
  ABC-I response is determined by ≥ 25% reduction in ABC-I score from baseline.
Change From Baseline on the ABC Subscale for Social Withdrawal at Week 8 | Week 8
Change From Baseline on the Stereotypic Behavior Subscale at Week 8 | Week 8
Change From Baseline on the Hyperactivity/Noncompliance Subscale at Week 8 | Week 8
Change From Baseline on the Inappropriate Speech Subscale at Week 8 | Week 8
Clinical Global Impression-Improvement (CGI-I) Score at Week 8 | Week 8
Number of Participants With Procholinergic Symptoms | Up to approximately 10 weeks
Number of Participants With Anticholinergic Symptoms | Up to approximately 10 weeks
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to approximately 10 weeks
Number of Participants With Serious Adverse Events (SAEs) | Up to approximately 10 weeks
Number of Participants With Adverse Events of Special Interest (AESIs) | Up to approximately 10 weeks
Number of Participants With AEs Leading to Discontinuation of Study Intervention | Up to approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (27):
  - Local Institution - 0036, Dothan, Alabama
  - Local Institution - 0236, Phoenix, Arizona
  - Local Institution - 0031, Anaheim, California
  - Local Institution - 0092, Chino, California
  - Local Institution - 0257, Glendale, California
  - Local Institution - 0181, San Rafael, California
  - Local Institution - 0252, Colorado Springs, Colorado
  - Local Institution - 0256, Hartford, Connecticut
  - Local Institution - 0264, Boca Raton, Florida
  - Local Institution - 0099, Gainesville, Florida
  - Local Institution - 0278, Gainesville, Florida
  - Local Institution - 0155, Peachtree Corners, Georgia
  - Local Institution - 0266, Chicago, Illinois
  - Local Institution - 0160, Bloomfield Hills, Michigan
  - Local Institution - 0220, Detroit, Michigan
  - Local Institution - 0110, Las Vegas, Nevada
  - Local Institution - 0246, Staten Island, New York
  - Local Institution - 0263, The Bronx, New York
  - Local Institution - 0247, West Chester, Ohio
  - Local Institution - 0269, Danville, Pennsylvania
  - Local Institution - 0105, Pittsburgh, Pennsylvania
  - Local Institution - 0041, Dallas, Texas
  - Local Institution - 0273, Fort Worth, Texas
  - Local Institution - 0185, Spring, Texas
  - Local Institution - 0074, Bountiful, Utah
  - Local Institution - 0271, Provo, Utah
  - Local Institution - 0260, Richmond, Virginia
- Argentina (6):
  - Local Institution - 0046, La Plata, Buenos Aires
  - Local Institution - 0048, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0047, Córdoba
  - Local Institution - 0288, Córdoba
  - Local Institution - 0049, Mendoza
  - Local Institution - 0140, Santiago del Estero
- Australia (4):
  - Local Institution - 0010, Westmead, New South Wales
  - Local Institution - 0007, Brisbane, Queensland
  - Local Institution - 0045, Melbourne, Victoria
  - Local Institution - 0286, Melbourne, Victoria
- Canada (5):
  - Local Institution - 0136, Edmonton, Alberta
  - Local Institution - 0134, Hamilton, Ontario
  - Local Institution - 0135, Kingston, Ontario
  - Local Institution - 0205, Toronto, Ontario
  - Local Institution - 0187, Montreal, Quebec
- India (3):
  - Local Institution - 0056, Kozhikode, Kerala
  - Local Institution - 0061, Nagpur, Maharashtra
  - Local Institution - 0218, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07284745.html